CLINICAL TRIAL: NCT02353637
Title: Partial Meal Replacements Providing High Protein, Restricted Carbohydrates in the Treatment of Adolescents With Severe Obesity: A Randomized Controlled Trial
Brief Title: The Peds Obesity Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Ideal PRotein of America (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UFJ 2014-140; IRB201702423 (Other: University of Florida)
Record Dates: First submitted 2015-01-21; First posted 2015-02-03 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Male High Protein, Restricted Carbo, Partial Meal Replacement (Active Comparator): A high protein, restricted carbohydrates diet that utilizes partial meal replacements
  Interventions: Dietary Supplement: Partial Meal Replacements
- Female High Protein, Restricted Carbo, Partial Meal Replaceme (Active Comparator): A high protein, restricted carbohydrates diet that utilizes partial meal replacements
  Interventions: Dietary Supplement: Partial Meal Replacements

INTERVENTIONS:
Dietary Supplement: Partial Meal Replacements — The use of partial meal replacements will be utilized in conjunction with a high protein, restricted carbohydrate diet

SUMMARY:
The aim of the study is to investigate, in severely obese adolescents, the effects of a high protein, restricted carbohydrates utilizing partial meal replacements diet (HPRC-PMR) on weight loss, body composition, and bio-chemical markers of lipid metabolism, insulin resistance, and inflammation over a 12 months period.

DETAILED DESCRIPTION:
Severely obese adolescents (13 to 17 year old males and post-menarcheal females between the ages of 12 and 17) will be recruited through the University of Florida Health Pediatric Weight Management Center. Therefore, all these patients would have undergone a multifaceted assessment that is part of the standard of care at the University of Florida Pediatric Weight Management Center. This includes a behavioral assessment conducted by the Center's psychologist, a detailed medical history and physical examination as well as a comprehensive laboratory testing to investigate for obesity comorbidities as indicated clinically for the individual patient. These laboratory tests include but not limited to the following: Complete Blood Count, comprehensive metabolic panel, liver enzymes, thyrotropin, fasting plasma glucose and insulin levels, fasting lipid profile and urinalysis. In addition, as part of the standard of care at the University of Florida Pediatric Weight Management Center, patients and families complete the Obesity and Quality of Life questionnaires as well as the University of Florida Pediatric Weight Management Center Physical Activity questionnaire. Inclusion criteria include adolescents with primary obesity and a BMI≥ 99th percentile for age. Exclusion criteria include current diagnosis of Type II Diabetes Mellitus; gall bladder, liver or renal disorders; known eating disorders; known endocrine disorders such as hypothyroidism or polycystic ovary syndrome; pregnancy; genetic disorder, such as Prader-Willi Syndrome; mental retardation; severe depression; or use of any chronic medication that could impact appetite significantly. Patients with poor family support that might potentially preclude compliance with the study requirements will also be excluded. These diseases will be ruled out by means of medical history, physical examination and standard of care laboratory tests obtained on patients upon their entry to the University of Florida Health Pediatric Weight Management Center. A urine pregnancy test will be performed on female adolescents prior to enrolment in the study. Written informed consent will be obtained from the parent and assent from the adolescent.

These patients will participate in a high protein, restricted carbohydrates utilizing partial meal replacements diet (HPRC-PMR) after obtaining consent to participate in the study.

Behavioral counseling will be provided to all participants in the study. The behavior modification used as part of the standard of care at the University of Florida Health Pediatric Weight Management Center includes a combination of immediate, short-term, and long-term individual and family psychotherapy sessions to increase motivation to change diet and physical activity level. These treatments may also help children cope with the emotional stresses associated with being overweight and boost confidence especially within the school system. Obesity and Quality of Life survey will be completed by patients at baseline, and at 3, 6 and 12 months after enrollment. (Permission to use this survey in the Center was obtained from Obesity and Quality of Life Consulting, Durham, North Carolina, and Children's Hospital Medical Center, OH). The survey includes questions regarding physical comfort, body esteem, social life and family relations.

Patients on the HPRC-PMR diet will follow 4 phases. Please see attached table for details.

The minimum amount of protein intake should be 1 g/Kg of protein/day. All meats and fish are permitted in this phase. Lean meats should be chosen. Patients will be encouraged to avoid hunger by having meals and 3 snacks throughout the day.

Enrolled participants will have scheduled meetings with the dietitian. The schedule involves weekly meetings for the first 2 months, then every other week for additional 4 months, followed by monthly meeting for additional 6 months for each patient/family.

Participants will be encouraged via the scheduled meetings with the dietitian to manage expected slip-ups. Minor, inconsequential slip-ups usually occur when the patient is not eating at home. In these cases, patients are encouraged to avoid carbohydrates, or starchy foods and desserts. In these cases, there will be no consequences, as long as these meals don't become a habit should go back to their regular diet the next day. A major diet slip-up is a big meal with all the trimmings. Patient will be encouraged to make up for a major diet slip-up the next day by avoiding all simple and complex carbohydrates for that one day only.

All participants will be encouraged to have "break day" in the maintenance phase. It is a day where the patient goes "all-out" and enjoys whatever foods they feel like eating! Dieters who have struggled with his/her weight and beef, poultry, pork or veal in place of the meal replacement at lunch.

ELIGIBILITY:
Inclusion Criteria:

* Severely obese adolescents (13 to 17 year old males and post-menarcheal females between the ages of 12 and 17) will be recruited through the UF Health Pediatric Weight Management Center.
* All patients would undergo a multifaceted assessment that is part of the standard of care at the UF Pediatric Weight Management Center. (This includes a behavioral assessment conducted by the Center's psychologist, a detailed medical history and physical examination as well as a comprehensive laboratory testing to investigate for obesity comorbidities as indicated clinically for the individual patient. These laboratory tests include but not limited to the following: CBC, comprehensive metabolic panel, liver enzymes, thyrotropin, fasting plasma glucose and insulin levels, fasting lipid profile and urinalysis.)
* As part of the standard of care at the UF Pediatric Weight Management Center, patients and families complete the IWQOL (Obesity and Quality of Life) questionnaires as well as the UF Pediatric Weight Management Center Physical Activity questionnaire.
* Adolescents with primary obesity and a BMI≥ 99th percentile for age.

Exclusion Criteria:

* Current Diagnosis of Type II Diabetes Mellitis
* Gall Bladder, Renal or Liver Disorders
* Known Eating Disorders
* Known Endocrine Disorders (such as hyperthyroidism or polycystic ovary syndrome)
* Pregnancy
* Genetic disorder (such as Prader-Willi Syndrome)
* Mental Retardation
* Severe Depression
* Use of any chronic medicine which could impact appetite

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Improvement in BMI-Z Scores | 12 months
  BMI measurements will be taken at all appointments for 12 months to track improvement in BMI
Weight Loss | 12 months
  Weigh will be obtained at each appointment to track weight loss of 12 months
Metabolic Abnormalities (Periodic labwork will be obtained over the 12 month period to monitor metabolic abnormalities) | 12 months
  Periodic labwork will be obtained over the 12 month period to monitor metabolic abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Madeline Joseph, MD, Principal Investigator — UFJP
Locations (1):
- University of Florida Pediatric Weight Management Center, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided